CLINICAL TRIAL: NCT01626287
Title: Reduction of Perineal Pain After Vaginal Birth With Black Tea: Pilot Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FHREB 2012-044
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2013-10

CONDITIONS: Perineal Pain
Keywords: perineal; postpartum; pain; treatment; ice and black tea; maternal satisfaction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Black tea bag (Experimental)
  Interventions: Other: Warm water soaked Black Tea Bags
- ice packs (Active Comparator): 20 randomly chosen participants will be given frozen ice packs for perineal pain relief
  Interventions: Other: Frozen perineal pad

INTERVENTIONS:
Other: Frozen perineal pad — Frozen ice pads will be provided as per participants' request
  Arms: ice packs
Other: Warm water soaked Black Tea Bags — warm water soaked black tea bags will be provided to participants' as per their request
  Arms: Black tea bag

SUMMARY:
Perineal trauma is common during vaginal birth. The discomfort this causes can interfere with a woman's recovery and early motherhood.Mothers are offered a standard treatment after childbirth, water soaked frozen peri pads (ice packs), to alleviate the discomfort. However, a Cochrane review questions the efficacy of ice packs treatment. An alternative treatment that may be more comfortable and effective for women is warm water soaked black tea bags. Medicinal use of black tea bags has been based on their astringent (shrinking or constricting) properties and have been used for various medical applications.

The investigators will conduct a pilot randomized controlled trial (RCT) of 40 pregnant mothers randomized to either intervention group (tea bags; n=20) or control group (ice packs; n=20). The goal of this pilot is to test the feasibility of a larger RCT by assessing recruitment, testing the protocol, and evaluating a proposed primary outcome objective of analgesic use during hospitalization as an indicator of pain. The investigators expect this pilot study to demonstrate feasibility for a large scale RCT to formally evaluate the efficacy of black tea bags to reduce perineal pain in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women (delivering their first baby) over the age of 19 who have delivered vaginally at Abbotsford Regional Hospital and Cancer Centre

Exclusion Criteria:

* multiparity (women who have delivered vaginally more than once), VBAC (Vaginal Birth after Cesarean Section), active sexually transmitted infection lesions, vulvar varicosities, third and forth degree perineal tear, hematoma, retained placenta/products, substance abuse, and other medical conditions requiring frequent analgesia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
use of analgesia during hospitalization | 24 hours post partum

CONTACTS AND LOCATIONS:
Overall Officials: Karmjit Kaur Sandhu, MScN, Principal Investigator — Fraser Health Authority
Locations (1):
- Abbotsford Regional Hospital and Cancer Centre, Abbotsford, British Columbia, Canada

REFERENCES:
- [Derived] East CE, Dorward ED, Whale RE, Liu J. Local cooling for relieving pain from perineal trauma sustained during childbirth. Cochrane Database Syst Rev. 2020 Oct 9;10(10):CD006304. doi: 10.1002/14651858.CD006304.pub4. PMID 33034900